CLINICAL TRIAL: NCT04558645
Title: Evaluation of Quality of Life, Physical Activity and Depression in Patients With Type 1 Diabetes Mellitus During the Covid-19 Pandemic
Brief Title: Evaluation of Quality of Life in Patients With Type 1 Diabetes Mellitus During the Covid-19 Pandemic
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Zeliha ÇELİK, Research assistant, Gazi University
Other Study IDs: 91610558-604.01.02
Record Dates: First submitted 2020-09-18; First posted 2020-09-22 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Type 1 Diabetes Mellitus; Covid19
MeSH Terms: conditions — Diabetes Mellitus, Type 1; COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with type 1 diabetes mellitus: Patients with Type 1 diabetes mellitus willing to participate in the study
  Interventions: Other: Online Survey
- Healthy controls: Healthy controls without chronic disease willing to participate in the study
  Interventions: Other: Online Survey

INTERVENTIONS:
Other: Online Survey — Online surveys will be applied to all participants

SUMMARY:
During the COVID-19 pandemic, the time spent at the home of patients has increased because of national quarantine policies and patients' fear of getting sick. For this reason, in this ongoing process, patients have been unable to go to work regularly due to their chronic diseases (being on administrative leave) and their fear of going out. These reasons have prevented being physically active. The aim of the study is to evaluate the physical activity level, quality of life, glucose control, anxiety, depression, fear of hypoglycemia and loneliness perceptions of patients with type 1 diabetes mellitus during the COVID-19 pandemic period and compared with healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with Type 1 Diabetes Mellitus
* Willing to participate in the study
* Participants whose native language is Turkish

Exclusion Criteria:

* Unwilling to participate in the study
* Having a cognitive disorder
* Not being literate
* Individuals who do not have sufficient knowledge and functional levels to fill out the online form

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with type 1 diabetes mellitus and healthy controls between 18-65 years
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2020-09-18 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2020-12-26 (Actual)

PRIMARY OUTCOMES:
Physical activity level | Five minutes
  Physical activity level using International Physical Activity Questionnaire - Short Form (IPAQ-SF) will be evaluated.
General Quality of life | Ten minutes
  Quality of life using Short Form Health Survey (SF-36) will be evaluated.

SECONDARY OUTCOMES:
Depression | Three minutes
  Depression using Hospital Anxiety and Depression Scale will be evaluated.
Anxiety | Three minutes
  Anxiety using Hospital Anxiety and Depression Scale will be evaluated.
Self-reported hypoglycemia | Last seven day
  It will be questioned how many times patients have had hypoglycemic attacks (<4 mmol/L and common symptoms) in the last 7 days.
Loneliness | Three minutes
  Loneliness using UCLA Loneliness Scale Short Form (ULS-8) will be evaluated.
Hypoglisemia fear | Five minutes
  Hypoglisemia fear using Hypoglisemia Fear Survey (HFS) will be evaluated.
Dyspnea | Two minutes
  Dyspnea during daily life activites using Modified Medical Research Dyspnea Scale will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Zeliha ÇELİK, MSc, Study Chair — Gazi University; Meral BOŞNAK GÜÇLÜ, Prof, Study Director — Gazi University; Füsun BALOŞ TÖRÜNER, Prof, Principal Investigator — Gazi University
Locations (1):
- Zeliha ÇELİK, Ankara, Çankaya, Turkey (Türkiye)